CLINICAL TRIAL: NCT01119157
Title: Comparison of the Cellular and the Humoral Immunogenicity as Well as the Safety of Different Trivalent Influenza Vaccines in Healthy Adults Between 18 and 60 Years of Age
Brief Title: Comparison of the Cellular and the Humoral Immunogenicity, Safety of Different Trivalent Influenza Vaccines
Acronym: FLUSECUOEKH1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Centre for Epidemiology, Hungary (Other Government)
Collaborators: Netherlands Vaccine Institute (Unknown); National Public Health Institute, Finland (Unknown)
Responsible Party: Dr Visontai Ildiko, National Centre for Epidemiology, Hungary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLUSECURE-OEK-H01; 2008-002307-22 (EudraCT Number)
Record Dates: First submitted 2010-05-04; First posted 2010-05-07 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Healthy Volunteers
Keywords: influenza vaccine; cellular immune response; humoral immune response
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; vaxigrip; influvac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- humoral and cellular immune response (Experimental)
  Interventions: Biological: influenza vaccine
- reactogenicity (Experimental)
  Interventions: Biological: influenza vaccine

INTERVENTIONS:
Biological: influenza vaccine — whole virus influenza vaccine adjuvanted with aluminium phosphate, 3 x 15 μg HA / 0.5 ml, for i.m. administration subunit influenza vaccine 3 x 15 μg HA / 0.5 ml, for i.m. administration split influenza vaccine 3 x 15 μg HA / 0.5 ml, for i.m. administration
  Other Names: FluvalAB adjuvanted trivalent seasonal influenza vaccine; Vaxigrip; Influvac

SUMMARY:
This is a randomized, single-blinded, Phase IV, monocentric study in healthy adults aged > 18 and < 60 years to evaluate the cellular and humoral immunogenicity as well as the reactogenicity of intramuscular, inactivated, trivalent influenza vaccines, including aluminium adjuvanted whole virus vaccine, split vaccine and subunit vaccine.

DETAILED DESCRIPTION:
This is a randomized, single-blinded study on vaccines for prevention of influenza.

Three study visits will be scheduled for each study subject, at Day 0, Day 9-11 and Day 30-35. Prior to the performance of any protocol procedures, the investigator is will obtain an informed consent from each participant.

At the first study visit (Day 0), demographic data, medical history, pre-existing conditions and concomitant medication will be recorded. Physical examination with recording of vital signs will be performed and in case of females of childbearing age, a pregnancy test will be performed. After the subject has qualified eligible, before vaccination, 60 ml venous blood will be taken for base-line immunity tests. Each subject will be randomly allocated to receive one of the three study vaccines, administered as a deep intramuscular (i.m.) injection into the deltoid muscle. The subjects will be blinded for the vaccine regimen. The principal investigator will administer the vaccines filled in ampoule or packed in pre-filled ready-to-use syringes and can thus not be blinded, but the staff and sub-investigators responsible for the routine follow-up and assessments and laboratory personnel will be blinded. A diary card will be given to each subject for recording pre-defined solicited adverse events for the vaccination day and 6 subsequent days and all other adverse events and concomitant medications.

At the second study visit (Day 9-11) the diary card will be collected. All adverse events and concomitant medication will be assessed and recorded. A physical examination will be performed and 60 ml venous blood shall be taken for immunity tests. A new diary card will be given to each subject for recording adverse events and concomitant medications.

At the third study visit (Day 30-35), the diary card will be collected. All adverse events and concomitant medication will be assessed and recorded. A physical examination will be performed and 60 ml venous blood shall be taken for immunity tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers > 18 and < 60 years of age, both sexes;
* Full contractual capacity of the participants
* Are in good health (as determined by vital signs and medical history);
* Negative urine or serum pregnancy test for females of childbearing potential.
* If the subject is female and of childbearing potential, she must use an acceptable contraception method and not become pregnant for the duration of the study. (Acceptable contraception includes implants, injectables, combined oral contraceptives, effective intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner);
* Are able to understand and comply with planned study procedures;
* Signed informed consent prior to initiation of study procedures;
* Absence of existence of any exclusion criteria

Exclusion Criteria:

* Known allergy to eggs OR other components of any of the vaccines (in particular mercury);
* History of Guillain-Barré syndrome;
* Pregnancy OR breast feeding OR positive pregnancy test prior to vaccination;
* Immunosuppressive therapy in the preceding 36 months;
* Active neoplasm (i.e. requiring any form of anti-neoplastic therapy);
* Concomitant corticosteroid therapy, including inhaled corticosteroids. Local corticosteroid or corticosteroid nasal spray are permitted.
* Psychiatric illness and/or concomitant psychiatric drug therapy that may have effect on full contractual capacity of the participant;
* Immunoglobulin (or similar blood product) therapy within 3 months prior to vaccination;
* Vaccine therapy within 4 weeks prior to the study;
* Influenza vaccination within 2 years prior to the study;
* Chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the immune response;
* Documented HIV, HBV or HCV infection;
* Acute febrile respiratory illness within one week prior to vaccination;
* Experimental drug therapy within 1 month prior to vaccination;
* Alcohol or drug abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Number of seroconversions, > 4-fold increase in Haemagglutination inhibition (HI), mean geometric increase and antibody titre the proportion of subjects achieving an HI titre > 40, virus neutralization assay, Granzyme B, INF-gamma, IL-10, side effects. | Day 35
  There remains substantial uncertainty about the clinical effectiveness of influenza vaccines based on current health care literature. The standard methodology to determine vaccine efficacy is based on hemagglutinin inhibition assay. Assays based on the immune response against the N antigen and based on the cellular immune response are now being designed and validated in the EU-funded Flusecure project. Importantly, recent EMEA regulations for registration of vaccines against avian influenza require an assessment of the cellular and the N-specific immune responses (EMEA/CHMP/VWP/263499/2006).

SECONDARY OUTCOMES:
Side effects | 65 days after vaccination
  In the course of tolerability assessment the frequency, mean time of appearance, duration and severity of the AEs (local and general) will be assessed according to CPMP/BWP/214/968: "Note for Guidance on Harmonization of Requirements for Influenza Vaccines", 12 March 1997, Para. 2.4., 2.6., and 3.2.

CONTACTS AND LOCATIONS:
Overall Officials: Ildikó Visontai, MD, Study Director — National Centre for Epidemiology
Locations (1):
- National Health Centre, Budapest, Hungary